CLINICAL TRIAL: NCT04701021
Title: Safety and Effect of Different Doses of TENDU Vaccine, a Therapeutic Peptide Conjugate Vaccine, in Patients With Relapse After Primary Radical Prostatectomy
Brief Title: TENDU Vaccine in Patients With Relapse After Primary Radical Prostatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ultimovacs ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TENDU-101
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
Keywords: prostate; vaccine; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENDU (Experimental): Three different doses of the TENDU vaccine are to be investigated: 40, 400 and 960μg.
  Interventions: Biological: TENDU

INTERVENTIONS:
Biological: TENDU — The vaccine is administrated by subcutaneous injections, one injection per drug substance (four separate injections) consecutively.

SUMMARY:
This is a phase I, dose selection study of safety and effect of different doses of TENDU vaccine, a therapeutic peptide conjugate vaccine, in patients with relapse after primary radical prostatectomy.

DETAILED DESCRIPTION:
This is a open label dose selection study to investigate the safety, tolerability, immune response and preliminary clinical effect of different doses of the TENDU vaccine. TENDU is a synthetic therapeutic peptide conjugate vaccine intended for treatment of prostate cancer.

The patients enrolled in this study is adults with documented progressive disease after radical prostatectomy and who are eligible for salvage radiotherapy and short-term (6 months) androgen deprivation therapy.

All patients taking part at the study must be vaccinated with a Boostrix vaccine (including tetanus antigen) one week prior to the first TENDU vaccine treatment.

Three different doses, 40, 400 and 960 μg of the TENDU vaccine are to be investigated.

The vaccine is administrated by subcutaneous injections with one injection per drug substance (four separate injections) consecutively. The TENDU vaccine will be given four times during a treatment period lasting for 6 weeks and followed up for 6 months after the last treatment.

In total between 12 to 18 patients will be enrolled with a 3+3 design in each dose cohort. The first patient will receive the lowest dose of the TENDU vaccine, and after the treatment is completed, a safety evaluation will be done to evaluate enrolment of the next patients in this cohort. If one patient develops a dose limiting toxicity at a specific dose, an additional three patients are to be enrolled into that same dose cohort, and on the recommended dose an addition of 3 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥18 years of age
2. PSA rise >0.2 ng/mL less than 18 months following radical prostatectomy (RP) and pathological ISUP Grade 4-5 (Gleason score >7), or persisting PSA >0.1 ng/mL six weeks after RP and short PSA-DT, eligible for salvage radiotherapy and short term androgen deprivation therapy
3. ECOG performance status 0 or 1
4. Adequate organ function as indicated by the following laboratory values:

   * White blood cell count ≥ 2,500/μL
   * Absolute neutrophil count ≥ 1,000/μL
   * Platelets ≥ 100,000/μL
   * Haemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
   * Serum total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN
   * AST and ALT ≤ 2.5 x ULN
5. Patients with potential to father children must use an acceptable contraceptive method
6. Written informed consent prior to any study-specific evaluations

Exclusion Criteria:

1. History of hematologic or primary solid tumor malignancy other than prostate cancer with remission less than 3 years prior study enrolment.
2. Metastatic disease assessed by PSMA PET/CT
3. Hypersensitivity to the active substance or any of its excipients
4. Current use of androgen deprivation therapy or radiotherapy to the pelvis
5. Known history or any evidence of active, non-infectious pneumonitis
6. History of New York Heart Association class 3-4 congestive heart failure or history of myocardial infarction within 6 months of starting study treatment
7. Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule.
8. Active infection requiring systemic therapy
9. Diagnosis of immunodeficiency
10. Any use of immunosuppressive (cytotoxic chemotherapy, systemic steroids) or immunomodulating agents within 8 weeks of study entry.
11. Hepatitis B or Hepatitis C or Human Immunodeficiency Virus positive
12. Expected to require any other form of systemic or localized antineoplastic therapy during the study
13. Received any other investigational therapy within 4 weeks of the first dose of study treatment
14. Any medical, psychological, social or neurological condition that would make it difficult for the patient to participate in the study and comply with the study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of TENDU vaccine | Time from enrollment until 6 months after last dose
  Frequency and severity of Adverse Events (AEs) graded according to CTCAE version 5.0.

SECONDARY OUTCOMES:
Assessment of Immunological response | Time from enrollment until 6 months after last dose
  To evaluate the immunological response against the prostate specific peptides in the patients at baseline and after TENDU vaccinations.
Assessment of anti-tetanus protein and anti-MTTE titers | Time from enrollment until 6 months after last dose
  To evaluate the preliminary anti-tumor activity of the TENDU vaccine in patients pre- and post the vaccination with Boostrix (including tetanus antigen) and the TENDU vaccinations by evaluation of anti-tetanus protein and anti-MTTE titers.
Assessment of Anti-tumor activity | Time from enrollment until 6 months after last dose
  To evaluate the preliminary anti-tumor activity of the TENDU vaccine according to changes in the PSA, PAP, PSMA and PET/CT.

OTHER OUTCOMES:
Assessment of antibody titers | Time from enrollment until 6 months after last dose
  Evaluation of antibody titers against PAP and PSMA peptides epitopes presented in the TENDU vaccine.
Assessment of possible biomarkers | Time from enrollment until 6 months after last dose
  Assessment of possible biomarkers e.g. phenotyping of circulating tumor cells (CTCs)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Lilleby, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, The Norwegian Radium Hospital, Oslo, Norway